CLINICAL TRIAL: NCT00894686
Title: Open-label Phase Iv Study To Investigate The Seropersistence Of Tick-borne Encephalitis (Tbe) Virus Antibodies After The First Booster And The Response To A Second Booster Vaccination With Fsme-immun In Children, Adolescents And Young Adults (Follow-up To Study 700401)
Brief Title: Tick-Borne Encephalitis (TBE) Seropersistence After First Booster and Response to a Second Booster in Children, Adolescents and Young Adults (Follow-Up to Study 700401)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Prevention
Other Study IDs: 700802; B9371021 (Other: Alias Study Number); 2009-009324-36 (EudraCT Number)
Record Dates: First submitted 2009-04-30; First posted 2009-05-07 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-05

CONDITIONS: Encephalitis, Tick-Borne
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental): Assessment of seropersistence of TBE antibodies at yearly intervals from approximately 3 years (38 months) to 10 years (118 months) after the first booster vaccination (in Study 700401), as well as antibody response to a second booster vaccination with either FSME-IMMUN 0.25 mL Junior or FSME-IMMUN 0.5 mL, depending on the subject´s age. Timing of the second booster vaccination will depend on the level of serum TBE antibodies detected at the defined assessment time points. Subjects who are not protected against TBE for an entire further season (NT titer <= 20 and/or ELISA value <=126 VIE U/mL) will be invited to receive the second booster vaccination at either the 40, 48, 60, 72, 84, 96, 108, or 120-month time point.
  Interventions: Biological: FSME-IMMUN 0.25 mL Junior (1.2 µg TBE antigen/0.25 mL) or FSME-IMMUN 0.5 mL (2.4µg TBE antigen/0.5 mL)

INTERVENTIONS:
Biological: FSME-IMMUN 0.25 mL Junior (1.2 µg TBE antigen/0.25 mL) or FSME-IMMUN 0.5 mL (2.4µg TBE antigen/0.5 mL) — Dosage form: solution/suspension; injectable. Dosage frequency: once. Mode of administration: intramuscular.

SUMMARY:
The main purpose of this study is to assess the seropersistence of TBE virus antibodies in children, adolescents and young adults who received the first booster vaccination with either FSME-IMMUN 0.25 mL Junior or FSME-IMMUN 0.5 mL in precursor Study 700401.

ELIGIBILITY:
Inclusion Criteria:

Subjects who participated in precursor Study 700401 and meet ALL of the following criteria are eligible for participation in this study:

* Subject / parent(s) / legal guardian(s) provide(s) written informed consent (according to national law);
* Subject provides written assent to the study according to age and capacity of understanding;
* Subject received the first booster vaccination with either FSME-IMMUN 0.25 ml Junior or FSME-IMMUN 0.5 ml during the course of precursor Study 700401;
* Blood was drawn after the first booster vaccination in precursor Study 700401;
* Subject / parent(s) / legal guardian(s) understand(s) the nature of the study and is / are willing to comply with the requirements of the protocol (e.g. return for follow-up visits, completion of the Subject Diary).

Exclusion Criteria:

Subjects who participated in precursor Study 700401 and meet ANY of the following criteria are not eligible for participation in this study:

* Subject received any TBE vaccination since his / her first booster vaccination in precursor Study 700401;
* Subject has a history of infection with or vaccination against other flaviviruses (e.g. Dengue fever, yellow fever, Japanese B encephalitis) since his / her first booster vaccination in precursor Study 700401;
* Subject is known to be HIV positive since his / her first booster vaccination in precursor Study 700401 (a special HIV test is not required for the purpose of the study);
* Subject received a blood product or immunoglobulins within 90 days before any blood draw or in the period between the blood draw and the booster vaccination (as applicable);
* Subject has a known or suspected problem with drug or alcohol abuse (> 4 liters of wine/week or equivalent level of other alcoholic beverages);
* Subject / parent(s) / legal guardian(s) is / are in a dependent relationship with the study investigator or with a study team member. Dependent relationship includes close relatives (i.e., children or grandchildren, partner / spouse, siblings) as well as employees of the investigator or the site conducting the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2009-04-26 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Eva-Maria Pöllabauer, MD, Study Director — Baxter Healthcare Corporation
Locations (4):
- Austria (2):
  - Grieskirchnerstr.17, Oberösterreich
  - Untergraben 2, Oberösterreich
- Dr. Ulrich Behre, Baden-Württemberg, Germany
- Niepubliczny Zakład Opieki Zdrowotnej Ośrodek Zdrowia w Lipsku, Zamość, Poland

REFERENCES:
- [Derived] Poellabauer E, Angermayr R, Behre U, Zhang P, Harper L, Schmitt HJ, Erber W. Seropersistence and booster response following vaccination with FSME-IMMUN in children, adolescents, and young adults. Vaccine. 2019 May 27;37(24):3241-3250. doi: 10.1016/j.vaccine.2019.03.032. Epub 2019 Mar 27. PMID 30928173
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=700802&StudyName=Open-label%20Phase%20Iv%20Study%20To%20Investigate%20The%20Seropersistence%20Of%20Tick-borne%20Encephalitis%20%28tbe%29%20Virus%20Antibodies%20After%20The%20First%20Booster%20And%20The%20Response%20To%20A%20Second%20Booster%20Vaccination%20With%20Fsme-immun%20In%20Children%2C%20Adolescents%20And%20Young%20Adults%20%28follow-up%20To%20Study%20700401%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a follow-up study of 700401 (NCT00161967) in which participants received the first booster vaccination.
Groups:
- FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL: Participants with low tick-borne encephalitis (TBE) serum antibody levels and received first booster vaccination in Study 700401 (NCT00161967) were administered single intramuscular injection of FSME-IMMUN 0.25 mL Junior (less than 16 years of age) or FSME-IMMUN 0.5 mL (16 years or above of age), as second booster vaccination in this study either at Month 40, 48, 60, 72, 84, 96, 108, or 120. Participants were followed up to 21-35 days post vaccination in this study.
Period: Overall Study
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Started | 179
Completed | 123
Not Completed | 56
Not completed — Withdrawal by Subject | 50
Not completed — Physician Decision | 1
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants enrolled into the study.
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 179
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 91
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 21-35 Days After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level greater than equal to (>=) 10 at 21-35 days after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent confidence interval (CI) was based upon the observed percentage of participants.
Time Frame: 21-35 days after first TBE booster vaccination
Population: Per-protocol population included participants who had been enrolled and meet all inclusion/exclusion criteria at all visits, had available assay results at any blood sampling visit and had no other major protocol deviation. Here, "Number of participants analyzed" (N) signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 171
Percentage of participants | 100.0 [97.9 to 100.0]

2. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 38 Months After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 38 months after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent confidence interval (CI) was based upon the observed percentage of participants.
Time Frame: 38 months after first TBE booster vaccination
Population: Per-protocol population included participants who had been enrolled and meet all inclusion/exclusion criteria at all visits, had available assay results at any blood sampling visit and had no other major protocol deviation. Here, "N" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 167
Percentage of participants | 100.0 [97.8 to 100.0]

3. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 46 Months After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 46 months after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 46 months after first TBE booster vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 147
Percentage of participants | 100.0 [97.5 to 100.0]

4. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 58 Months After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 58 months after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 58 months after first TBE booster vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 156
Percentage of participants | 99.4 [96.5 to 100.0]

5. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 70 Months After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 70 months after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 70 months after first TBE booster vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 157
Percentage of participants | 98.1 [94.5 to 99.6]

6. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 82 Months After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 82 months after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 82 months after first TBE booster vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 156
Percentage of participants | 96.8 [92.7 to 99.0]

7. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 94 Months After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 94 months after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 94 months after first TBE booster vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 156
Percentage of participants | 95.5 [91.0 to 98.2]

8. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 106 Months After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 106 months after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 106 months after first TBE booster vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 156
Percentage of participants | 94.9 [90.1 to 97.8]

9. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 118 Months After the First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 118 months after the first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 118 months after first TBE booster vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 155
Percentage of participants | 90.3 [84.5 to 94.5]

10. Primary Outcome: Seropositivity Rate Measured by Neutralization Test (NT) at 21-35 Days After the Second Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700802
Description: Seropositivity rate was reported as percentage of participants with NT level >=10 at 21-35 days after the second TBE booster vaccination. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 21-35 days after second TBE booster vaccination
Population: Per-protocol population included participants who had been enrolled and meet all inclusion/exclusion criteria at all visits, had available assay results at any blood sampling visit and had no other major protocol deviation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 26
Percentage of participants | 100.0 [86.8 to 100.0]

11. Secondary Outcome: Seropositivity Rate Measured by Enzyme-Linked Immunosorbent Assay (ELISA) at Each Available Time Point After First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Seropositivity rate was reported as percentage of participants with ELISA level greater than (>) 126 vienna units per milliliter (VIE U/mL) at each blood sampling time point after first TBE booster vaccination in Study 700401. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 21-35 days and 38, 46, 58, 70, 82, 94, 106, 118 months after first TBE booster vaccination
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 172
Percentage of participants
  After 21-35 days: number analyzed (Participants) | 171
  After 21-35 days | 98.8 [95.8 to 99.9]
  After 38 months: number analyzed (Participants) | 166
  After 38 months | 97.0 [93.1 to 99.0]
  After 46 months: number analyzed (Participants) | 146
  After 46 months | 100.0 [97.5 to 100.0]
  After 58 months: number analyzed (Participants) | 157
  After 58 months | 97.5 [93.6 to 99.3]
  After 70 months: number analyzed (Participants) | 156
  After 70 months | 96.8 [92.7 to 99.0]
  After 82 months: number analyzed (Participants) | 156
  After 82 months | 96.2 [91.8 to 98.6]
  After 94 months: number analyzed (Participants) | 156
  After 94 months | 96.2 [91.8 to 98.6]
  After 106 months: number analyzed (Participants) | 156
  After 106 months | 91.7 [86.2 to 95.5]
  After 118 months: number analyzed (Participants) | 155
  After 118 months | 87.7 [81.5 to 92.5]

12. Secondary Outcome: Seropositivity Rate Measured by Enzyme-Linked Immunosorbent Assay (ELISA) at 21-35 Days After Second Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700802
Description: Seropositivity rate was reported as percentage of participants with ELISA level >126 VIE U/mL at 21-35 days after second TBE booster vaccination. Exact 2-sided 95 percent CI was based upon the observed percentage of participants.
Time Frame: 21-35 days after second TBE booster vaccination
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 26
Percentage of participants | 100.0 [86.8 to 100.0]

13. Secondary Outcome: Geometric Mean Concentration Measured by Enzyme-linked Immunosorbent Assay (ELISA) at Each Available Time-Point After First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Antibody against TBE booster vaccination was measured as geometric mean concentration (GMC) by ELISA level at different time points after first booster vaccination. CIs were computed by back transforming the CIs based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 21-35 days and 38, 46, 58, 70, 82, 94, 106, 118 months after first TBE booster vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: VIE U/mL
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 172
VIE U/mL
  After 21-35 days: number analyzed (Participants) | 171
  After 21-35 days | 4368.2 [3605.22 to 5292.63]
  After 38 months: number analyzed (Participants) | 166
  After 38 months | 1081.5 [933.04 to 1253.51]
  After 46 months: number analyzed (Participants) | 146
  After 46 months | 1212.1 [1055.77 to 1391.65]
  After 58 months: number analyzed (Participants) | 157
  After 58 months | 1005.1 [876.16 to 1153.08]
  After 70 months: number analyzed (Participants) | 156
  After 70 months | 883.4 [767.09 to 1017.25]
  After 82 months: number analyzed (Participants) | 156
  After 82 months | 728.6 [626.66 to 847.12]
  After 94 months: number analyzed (Participants) | 156
  After 94 months | 636.8 [541.70 to 748.55]
  After 106 months: number analyzed (Participants) | 156
  After 106 months | 561.0 [469.95 to 669.58]
  After 118 months: number analyzed (Participants) | 155
  After 118 months | 506.4 [414.96 to 618.10]

14. Secondary Outcome: Geometric Mean Concentration Measured by Enzyme-linked Immunosorbent Assay (ELISA) at 21-35 Days After Second Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700802
Description: Antibody against TBE booster vaccination was measured as GMC by ELISA level after the second booster vaccination. CIs were computed by back transforming the CIs based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: 21-35 days after second TBE booster vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: VIE U/mL
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 26
VIE U/mL | 1844.1 [1305.54 to 2604.91]

15. Secondary Outcome: Geometric Mean Titer Measured by Neutralization Test (NT) Each Available Time-Point Blood Draw After First Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700401
Description: Antibody against TBE booster vaccination was measured as geometric mean titer (GMT) by NT level at different time points after first booster vaccination. CIs were computed by back transforming the CIs based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 21-35 days and 38, 46, 58, 70, 82, 94, 106, 118 months after first TBE booster vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 172
Titers
  After 21-35 days: number analyzed (Participants) | 171
  After 21-35 days | 380.7 [336.73 to 430.31]
  After 38 months: number analyzed (Participants) | 167
  After 38 months | 162.1 [139.29 to 188.58]
  After 46 months: number analyzed (Participants) | 147
  After 46 months | 108.1 [92.41 to 126.34]
  After 58 months: number analyzed (Participants) | 156
  After 58 months | 111.3 [96.10 to 128.84]
  After 70 months: number analyzed (Participants) | 157
  After 70 months | 123.4 [105.31 to 144.59]
  After 82 months: number analyzed (Participants) | 156
  After 82 months | 122.3 [102.33 to 146.28]
  After 94 months: number analyzed (Participants) | 156
  After 94 months | 82.8 [68.88 to 99.57]
  After 106 months: number analyzed (Participants) | 156
  After 106 months | 56.0 [46.42 to 67.57]
  After 118 months: number analyzed (Participants) | 155
  After 118 months | 53.9 [43.40 to 66.87]

16. Secondary Outcome: Geometric Mean Titer Measured by Neutralization Test (NT) After Second Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700802
Description: Antibody against TBE booster vaccination was measured as GMT by NT level after second booster vaccination. CIs were computed by back transforming the CIs based on the Student t distribution for the mean logarithm of the titers.
Time Frame: 21-35 days after second TBE booster vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 26
Titers | 126.8 [94.76 to 169.64]

17. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Antibody Concentrations After Second Tick-borne Encephalitis (TBE) Booster Vaccination as Compared to Before the Booster Vaccination as Measured by Enzyme-Linked Immunosorbent Assay (ELISA)
Description: GMFR in antibody concentration from pre-booster (before second booster vaccination) to post-booster (21-35 days after TBE vaccination) was measured by ELISA. CIs were computed by back transforming the CIs based on the Student t distribution for the mean logarithm of the titers, concentrations or the fold rises.
Time Frame: Before second booster vaccination (pre-vaccination), 21-35 days after second booster vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 26
Fold rise | 8.6 [6.69 to 11.10]

18. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Antibody Titer After Second Tick-borne Encephalitis (TBE) Booster Vaccination as Compared to Before the Booster Vaccination as Measured by Neutralization Test (NT)
Description: GMFR in antibody titers from pre-booster (before second booster vaccination) to post-booster (21-35 days after TBE vaccination) was measured by ELISA. CIs were computed by back transforming the CIs based on the Student t distribution for the mean logarithm of the titers, concentrations or the fold rises.
Time Frame: Before second booster vaccination (pre-vaccination), 21-35 days after second booster vaccination
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 26
Fold rise | 5.2 [2.78 to 9.67]

19. Secondary Outcome: Number of Participants With Injection Site Reactions and Systemic Reactions After Second Tick-borne Encephalitis (TBE) Booster Vaccination in Study 700802
Description: Injection site reactions included swelling, induration, redness, injection site pain, tenderness, ecchymosis and hematoma. Systemic reaction included headache, nausea, vomiting, muscle pain, joint pain, swelling of the lymph nodes, malaise and fatigue. Participants with any injection site reaction and systemic reaction after second TBE booster vaccination in Study 700802 were reported in this outcome measure.
Time Frame: From second booster vaccination up to 21-35 days after the vaccination
Population: The safety population included any participant who had received the second booster dose.
Measure: Number; unit: Participants
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
Number analyzed (Participants) | 26
Participants
  Injection site reactions | 1
  Systemic reactions | 0

ADVERSE EVENTS:
Time Frame: From second booster vaccination up to 21-35 days after the vaccination
Description: The safety population included any participant who had received the second booster dose.
Arm/Group | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSME-IMMUN 0.25 Milliliters (mL) Junior/0.5 mL (N=26)
Tenderness (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-06-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT00894686/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT00894686/SAP_001.pdf